CLINICAL TRIAL: NCT02101827
Title: Safety and Efficacy of Distending Media Infusion by Manual Syringe Method for Hysteroscopic Procedures
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 103006-E
Record Dates: First submitted 2014-03-06; First posted 2014-04-02 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Hysteroscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Hysteroscopic surgery: Women who received hysteroscopic surgeries or examinations

SUMMARY:
To evaluate the safety and efficacy of manual syringe-infusion method in hysteroscopic procedures.

DETAILED DESCRIPTION:
In order to minimize the amount of distending media infused during hysteroscopic procedures, investigators used manual syringe method for delivering of distending media during hysteroscopic procedures from June 2010 to November 2013 in our institute. The aim of this study was to evaluate the safety and efficacy of manual syringe-infusion method in hysteroscopic procedures.

The medical records of all women who received hysteroscopic procedures by manual fluid-infusion method or convention pump fluid infusion method between June 2010 and November 2013 will be reviewed. In order to reveal the superiority/inferiority of clinical outcome of women receiving manual fluid infusion method, perioperative outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Of greater than twenty-year-old female patients suffering from abnormal uterine bleeding, suspected endometrial lesions, endometrial polyp, or submucous myoma.
* Patients had hysteroscopic procedures for either diagnostic or therapeutic purpose from June 2010 to November 2013 in Department of Obstetrics & Gynecology in Far Eastern Memorial Hospital.

Exclusion Criteria:

* Female patients of less than twenty years-old.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had hysteroscopic procedures for either diagnostic or therapeutic purpose
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety of manual fluid-distension methods for hysteroscopic procedures | 1 week
  The complications (such as hyponatremia, abdominal pain) related to manual fluid-distension methods for hysteroscopic procedures.

SECONDARY OUTCOMES:
Feasibility of manual fluid-infusion methods for hysteroscopic procedures | 1 week
  The perioperative data, including operation time, estimated blood loss, completion operation rate of hysteroscopic procedure by using manual fluid-infusion methods

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan